CLINICAL TRIAL: NCT01725217
Title: A Phase 3, Multi-center, Open-label Study to Evaluate Immunogenicity and Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) in Healthy Children, Adolescents and Adults in Russia
Brief Title: Immunogenicity and Safety of Meningococcal ACWY Conjugate Vaccine in Healthy Children, Adolescents and Adults in Russia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V59_50
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Meningococcal Disease
Keywords: Meningitis; children; adolescents; adults; MenACWY
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MenACWY-CRM (Experimental): MenACWY-CRM
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — 1 vaccination at visit 1, conjugate vaccine, Intramuscular (IM) injection

SUMMARY:
To evaluate the immune response and safety following a single dose of Novartis Meningococcal ACWY conjugate vaccine (MenACWY-CRM) in healthy children, adolescents and adults in Russia.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment in this study were those:

1. Who were of any gender, from the age of 2 years and above at the time of visit 1, and to whom the nature of the study had been described and:

   * the parent/legal representative had provided written informed consent (≥2 to <18 years of age),
   * had provided written assent (≥11 to <18 years of age),
   * had provided written informed consent (≥18 years of age onwards).
2. Who the investigator believed that the subject and/or his or her parent/legal representative could and would comply with the requirements of the protocol (e.g., completion of the Diary Card, return for follow-up visit).
3. Who were in good health as determined by

   * medical history
   * physical exam
   * clinical judgment of the investigator
4. Who had a negative urine pregnancy test for female subjects from 11 years of age.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study were those:

1. Who were unwilling or unable to give written informed assent or consent to participate in the study.
2. Who were perceived to be unreliable or unavailable for the duration of the study period.
3. Who had a previous confirmed or suspected disease caused by N meningitidis.
4. Who had household contact with and/or intimate exposure to an individual with culture-proven N meningitidis infection within 60 days prior to enrollment.
5. Who had previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational).
6. Who were pregnant or breast feeding (female subjects).
7. Who had received any investigational or non-registered product (drug or vaccine) within 28 days prior to enrollment or who expected to receive an investigational drug or vaccine prior to the completion of the study.
8. Who had received any vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who were planning to receive any vaccine within 30 days from the study vaccines.

   (Exception: Influenza vaccine might be administered up to 15 days prior to study vaccination and at least 15 days after study vaccination).
9. Who had experienced within the 7 days prior to enrollment significant acute infection (for example requiring systemic antibiotic treatment or antiviral therapy) or had experienced fever (defined as body temperature ≥ 38°C) within 3 days prior to enrollment.
10. Who had any serious acute, chronic or progressive disease (e.g., any history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), or blood dyscrasias, with signs of cardiac or renal failure or severe malnutrition). Who had epilepsy or any progressive neurological disease or history of Guillain-Barre syndrome.
11. Who had a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components including diphtheria toxin (CRM-197) and latex in the syringe.
12. Who had a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * receipt of immunosuppressive therapy within 30 days prior to enrollment (any systemic corticosteroid administered for more than 5 days, or in a daily dose > 1 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy)
    * receipt of immunostimulants
    * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study
13. Who were known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (4):
- Russia (4):
  - Federal State Budgetary Institution 'State Scientific Center 'Institution of Immunology' of the Russian Federal Biomedical Agency', Kashirskoye Highway, Moscow
  - Institution of the Russian Academy of Sciences "Scientific Center for Children Health RAMS", Lomonosovskiy Avenue, Moscow
  - Federal Budgetary Institution of Science 'St-Petersburg Scientific-Research Institution of Epidemiology and Microbiology by name of Pasteur', Mira Street, Sankt-Peterburg
  - Federal State Institution 'Scientific-Research Institution of Children's Infections of the Russian Federal Biomedical Agency', Prof.Popova Street, Sankt-Peterburg

REFERENCES:
- [Background] Trotter CL, Andrews NJ, Kaczmarski EB, Miller E, Ramsay ME. Effectiveness of meningococcal serogroup C conjugate vaccine 4 years after introduction. Lancet. 2004 Jul 24-30;364(9431):365-7. doi: 10.1016/S0140-6736(04)16725-1. PMID 15276396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 5 centers in Russia
Pre-assignment Details: All enrolled subjects were included in the study
Groups:
- ≥2 to ≤10 Years: Subjects ≥2 to ≤10 years of age who received one vaccination of MenACWY-CRM
- ≥11 to ≤17 Years: Subjects ≥11 to ≤17 years of age who received one vaccination of MenACWY-CRM
- ≥18 Years: Subjects ≥18 years of age who received one vaccination of MenACWY-CRM
Period: Overall Study
Arm/Group | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Started | 66 | 66 | 66
Completed | 65 | 66 | 66
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years | Total
Number analyzed (Participants) | 66 | 66 | 66 | 198
Age, Continuous [Mean (Standard Deviation); unit: year] | 6.0 (2.7) | 13.8 (2.1) | 38.8 (12.5) | 19.6 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 35 | 29 | 44 | 108
  MALE | 31 | 37 | 22 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Overall Subjects With Seroresponse After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as the percentages of overall subjects with hSBA (human serum bactericidal assay) seroresponse, directed against Neisseria meningitidis (N meningitidis) serogroups A, C, W and Y, 28 days after one vaccination of MenACWY-CRM (day 29).
  The seroresponse is defined as the percentages of subjects achieving hSBA ≥1:8 postvaccination with a prevaccination hSBA <1:4 and the percentages of subjects achieving at least four-fold increases in postvaccination hSBA from day 1 in subjects with a baseline hSBA ≥1:4
Time Frame: Day 29
Population: Analysis was done on Full Analysis Set (FAS), i.e., all subjects in the exposed population who provided one evaluable serum sample whose assay result is available for at least one serogroup at baseline and at day 29
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Overall (≥2 Years): All subjects ≥2 years of age who received one vaccination of MenACWY-CRM
Arm/Group | Overall (≥2 Years)
Number analyzed (Participants) | 193
Percentage of subjects
  MenA | 85 [79 to 90]
  MenC | 74 [67 to 80]
  MenW | 60 [53 to 67]
  MenY | 83 [77 to 88]

2. Secondary Outcome: Percentages of Subjects With Seroresponse After MenACWY-CRM Vaccination, by Age Group
Description: Immunogenicity was measured as the percentages of subjects stratified by age group with hSBA response, directed against N meningitidis serogroups A, C, W and Y, 28 days after one vaccination of MenACWY-CRM
Time Frame: Day 29
Population: Analysis was done on FAS dataset
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Number analyzed (Participants) | 63 | 65 | 65
Percentage of subjects
  MenA | 89 [78 to 95] | 89 [79 to 96] | 77 [65 to 86]
  MenC | 69 [56 to 80] | 82 [70 to 90] | 71 [58 to 81]
  MenW | 73 [60 to 83] | 51 [38 to 63] | 57 [44 to 69]
  MenY | 77 [65 to 87] | 88 [77 to 95] | 85 [74 to 92]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Subjects at Baseline and After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as hSBA GMTs, against N meningitidis serogroups A, C, W and Y, at baseline (day 1) and 28 days after MenACWY-CRM vaccination (day 29), overall and by age group
Time Frame: Days 1 and 29
Population: Analysis was done on FAS dataset
Measure: Geometric Mean (95% Confidence Interval); unit: human serum bactericidal assay titer
Arm/Group | Overall (≥2 Years) | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Number analyzed (Participants) | 193 | 63 | 65 | 65
human serum bactericidal assay titer
  MenA (Day 1) | 2.35 [2.17 to 2.55] | 2.17 [1.79 to 2.62] | 2.43 [2.01 to 2.93] | 2.61 [2.11 to 3.23]
  MenA (Day 29) | 93 [73 to 119] | 67 [38 to 119] | 134 [77 to 233] | 76 [41 to 143]
  MenC (Day 1) | 4.07 [3.45 to 4.8] | 3.16 [2.18 to 4.57] | 3.59 [2.5 to 5.15] | 6.68 [4.43 to 10]
  MenC (Day 29) | 59 [43 to 81] | 28 [14 to 56] | 47 [24 to 92] | 112 [52 to 243]
  MenW (Day 1) | 12 [9.42 to 15] | 7.93 [4.69 to 13] | 21 [13 to 36] | 13 [7.16 to 23]
  MenW (Day 29) | 111 [89 to 139] | 94 [56 to 155] | 117 [72 to 191] | 143 [83 to 248]
  MenY (Day 1) | 2.93 [2.61 to 3.28] | 3.02 [2.33 to 3.92] | 3.73 [2.89 to 4.82] | 2.74 [2.05 to 3.66]
  MenY (Day 29) | 58 [46 to 74] | 32 [18 to 56] | 67 [39 to 115] | 80 [43 to 147]

4. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥1:8 at Baseline and After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as the percentages of subjects with hSBA titer ≥1:8, at baseline (day 1) and 28 days after MenACWY-CRM vaccination (day 29), overall and by age group
Time Frame: Days 1 and 29
Population: Analysis was done on FAS dataset
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Overall (≥2 Years) | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Number analyzed (Participants) | 193 | 63 | 65 | 65
Percentage of Subjects
  MenA (Day 1) | 6 [3 to 10] | 2 [0.04 to 9] | 5 [1 to 13] | 11 [4 to 21]
  MenA (Day 29) | 89 [83 to 93] | 89 [78 to 95] | 92 [83 to 97] | 85 [74 to 92]
  MenC (Day 1) | 26 [20 to 33] | 13 [6 to 23] | 17 [9 to 28] | 49 [37 to 62]
  MenC (Day 29) | 84 [78 to 89] | 76 [63 to 86] | 86 [75 to 93] | 89 [79 to 96]
  MenW (Day 1) | 57 [50 to 64] | 30 [19 to 43] | 71 [58 to 81] | 69 [57 to 80]
  MenW (Day 29) | 97 [93 to 99] | 95 [87 to 99] | 98 [92 to 100] | 97 [89 to 100]
  MenY (Day 1) | 16 [11 to 22] | 10 [4 to 20] | 15 [8 to 26] | 22 [12 to 33]
  MenY (Day 29) | 88 [82 to 92] | 79 [67 to 88] | 94 [85 to 98] | 89 [79 to 96]

5. Secondary Outcome: Percentages of Subjects Aged 2 Through 5 Years With Solicited Local and Systemic AEs After MenACWY-CRM Vaccination
Description: Safety was assessed as the percentages of subjects aged 2 through 5 years who reported solicited local and systemic AEs within days 1 through 7 after MenACWY-CRM vaccination
Time Frame: Within days 1 through 7 postvaccination
Population: Analysis was done on safety dataset, i.e. all subjects in the exposed population who provided any post-baseline safety data
Measure: Number; unit: Percentage of subjects
Groups:
- ≥2 to ≤5 Years: Subjects ≥2 to ≤5 years of age who received one vaccination of MenACWY-CRM
- ≥2 to ≤3 Years: Subjects ≥2 to ≤3 years of age who received one vaccination of MenACWY-CRM
Arm/Group | ≥2 to ≤5 Years | ≥2 to ≤3 Years
Number analyzed (Participants) | 27 | 18
Percentage of subjects
  Tenderness | 41 | 39
  Erythema | 26 | 28
  Induration | 19 | 17
  Change in Eating Habits | 4 | 6
  Sleepiness | 33 | 28
  Irritability | 26 | 17
  Vomiting | 4 | 0
  Diarrhea | 11 | 11
  Rash | 4 | 6
  Fever (≥38 °C) | 4 | 6
  Use of analgesics/antipyretics | 7 | 0

6. Secondary Outcome: Percentages of Subjects Aged ≥6 Years With Solicited Local and Systemic AEs After MenACWY-CRM Vaccination
Description: Safety was assessed as the percentages of subjects aged ≥6 years who reported solicited local and systemic AEs within days 1 through 7 after MenACWY-CRM vaccination, overall and by age group
Time Frame: Within days 1 through 7 postvaccination
Population: Analysis was done on safety dataset
Measure: Number; unit: Percentage of Subjects
Groups:
- Overall (≥6 Years): All subjects ≥6 years of age who received one vaccination of MenACWY-CRM
- ≥6 to ≤10 Years: Subjects ≥6 to ≤10 years of age who received one vaccination of MenACWY-CRM
Arm/Group | Overall (≥6 Years) | ≥6 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Number analyzed (Participants) | 170 | 38 | 66 | 66
Percentage of Subjects
  Pain | 48 | 42 | 50 | 50
  Erythema | 18 | 18 | 18 | 17
  Induration | 14 | 11 | 17 | 12
  Chills | 9 | 8 | 8 | 12
  Nausea | 8 | 3 | 11 | 8
  Malaise | 20 | 16 | 23 | 20
  Myalgia | 19 | 13 | 29 | 14
  Arthralgia | 9 | 3 | 11 | 11
  Headache | 25 | 18 | 27 | 27
  Rash | 2 | 3 | 0 | 5
  Fever (≥38 °C) | 3 | 5 | 3 | 2
  Use of analgesic/antipyretics | 11 | 18 | 9 | 9

7. Secondary Outcome: Percentages of Subjects Reporting Unsolicited Adverse Events (AEs) After MenACWY-CRM Vaccination
Description: Safety was assessed in terms of percentages of subjects who reported all the adverse events (AEs) occurring from day 1 through 7, medically attended AEs, SAEs and AEs resulting in premature withdrawal, from day 1 through 29, after MenACWY-CRM vaccination, overall and by age group
Time Frame: AEs occurring from day 1 through 7, medically attended AEs, SAEs and AEs resulting in premature withdrawal, from day 1 through 29
Population: Analysis was done on safety dataset
Measure: Number; unit: percentage of subjects
Arm/Group | Overall (≥2 Years) | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years
Number analyzed (Participants) | 197 | 65 | 66 | 66
percentage of subjects
  Any AEs(days 1 through 7) | 17 | 20 | 12 | 18
  At least possibly related AEs (days 1 through 7) | 10 | 3 | 9 | 18
  SAE(days 1 through 29) | 0 | 0 | 0 | 0
  At least possibly related SAE(days 1 through 29) | 0 | 0 | 0 | 0
  Medically attended AE(days 1 through 29) | 4 | 8 | 2 | 3
  Premature withdrawal due to AE(days 1 through 29) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From day 1 through day 29
Description: Serious adverse events (SAEs) were collected from day 1 through day 29
Arm/Group | ≥2 to ≤10 Years | ≥11 to ≤17 Years | ≥18 Years | Overall (≥2 Years)
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 0/66 | 0/197
Other Adverse Events (participants affected / at risk) | 42/65 | 42/66 | 44/66 | 128/197
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ≥2 to ≤10 Years (N=65) | ≥11 to ≤17 Years (N=66) | ≥18 Years (N=66) | Overall (≥2 Years) (N=197)
Nausea (Gastrointestinal disorders) | 1 | 7 | 5 | 13
Chills (General disorders) | 3 | 5 | 8 | 16
Injection site erythema (General disorders) | 12 | 13 | 10 | 35
Injection site induration (General disorders) | 8 | 11 | 8 | 27
Injection site pain (General disorders) | 27 | 33 | 33 | 93
Irritability (General disorders) | 7 | 0 | 0 | 7
Malaise (General disorders) | 6 | 15 | 13 | 34
Rhinitis (Infections and infestations) | 6 | 0 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7 | 7 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 19 | 9 | 33
Headache (Nervous system disorders) | 8 | 18 | 18 | 44
Somnolence (Nervous system disorders) | 9 | 1 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less